CLINICAL TRIAL: NCT01140230
Title: Structural and Clinical Outcomes After Repair of Acute Rotator Cuff Tears
Brief Title: Outcomes After Repair of Acute Rotator Cuff Tears
Acronym: HBStud2
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: MD. Andreas Meunir, Department of Orthopeadic, Linkoeping University Hospital
Other Study IDs: Hanna Björnsson study 2
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2009-09

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; rotator cuff repair; age; timing to surgery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Few studies are considering acute traumatic rotator cuff tears in previously asymptomatic patients. The purpose of the current study was to investigate if delay of surgery, age at repair and the number of cuff tendons involved affected the structural and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* significant trauma to the shoulder
* sudden onset of symptoms
* asymptomatic in the shoulder before trauma
* pseudoparalysis in the shoulder after trauma
* full thickness rotator cuff tear of at least one tendon

Exclusion Criteria:

* patients with previous or gradual onset of symptoms in the traumatised shoulder
* partial rotator cuff tear
* displaced fracture

Ages: 42 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective review of our computerized database identified 49 patients repaired at our institution between May 2004 until May 2009 due to acute traumatic rotator cuff tears. 42 patients who fulfilled the inclusion criteria, were willing to participate in a follow-up evaluation after written and oral informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Adolfsson, Associate Professor, Study Director — Department of Orthopeadic, Linkoeping University Hospital

REFERENCES:
- [Background] Bassett RW, Cofield RH. Acute tears of the rotator cuff. The timing of surgical repair. Clin Orthop Relat Res. 1983 May;(175):18-24. PMID 6839586
- [Background] Lahteenmaki R, Lawrence S. Public biotech 2006 - the numbers. Nat Biotechnol. 2007 Jul;25(7):729-37. doi: 10.1038/nbt0707-729. No abstract available. PMID 17621294